CLINICAL TRIAL: NCT04689373
Title: Physical and Cognitive Effects of Fluoroscopy on Medical Professionals in the Operating Room : A Prospective Observational Study
Brief Title: Physical and Cognitive Effects of Fluoroscopy
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator, M.D., Istanbul University
Other Study IDs: 2020/1424
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Dehydration; Radiation Exposure
Keywords: medical professionals; intraoperative fluoroscopy; low dose radiation
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: VAS Score — The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.
  The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills.
  Other Names: Mini Mental State Examination

SUMMARY:
Background and objectives:

The researchers will perform this study to reveal the clinical meaning of fatigue, headache, diarrhea, and impaired cognitive functions that are often expressed verbally in healthcare professionals who are exposed to fluoroscopy.

Methods:

After obtaining written informed consent, 84 samples will be included in the study. For operating room employees who meet the criteria determined before and after the operation; mini-mental state examination, weight, heart rate, non-invasive blood pressure value, VAS score for headache, radiation exposure time on fluoroscopy device, Rad measurement with the help of personal dosimeter before and after surgery, and total time in the operating room will be recorded.

DETAILED DESCRIPTION:
Background and objectives:

Nowadays, operations under fluoroscopy are performed at increasing rates with the aim of increasing case management and surgical success. Due to this increasing exposure to radiation, it is important to show that fluoroscopy has an impact on employees not only annually but also daily. The researchers will perform this study to reveal the clinical meaning of fatigue, headache, diarrhea, and impaired cognitive functions that are often expressed verbally in healthcare workers who are exposed to fluoroscopy.

Methods:

After obtaining written informed consent; 84 samples consisting of orthopedic surgery and anesthesia residents and orthopedic operating room nurses between the ages of 18-60 who do not have cardiological, neurological and psychiatric diseases, have had fluoroscopic operations lasting more than 2 hours, wear protective scopy gowns and collar during surgery, will be included in the study. The total number of samples required for the study will be reached by taking repeated measurements on consecutive days from the same sample group, but not on the same day. For operating room employees who meet the criteria determined before and after the operation; mini-mental state examination, weight, heart rate, non-invasive blood pressure value, VAS score for headache, radiation exposure time on fluoroscopy device, Rad measurement with the help of personal dosimeter before and after surgery, and total time in the operating room will be recorded. This prospective study will be executed between December 2020 and June 2021.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study
2. ASA classification 1 or 2
3. Not leaving the operating room during the operation
4. To be carrying a fluoroscopy gown, protective collar, and dosimeter.

Exclusion Criteria:

1. Having a psychiatric illness
2. Having a neurological disease
3. Being under the age of 18
4. Presence of cardiac pathology
5. Being pregnant or suspected of pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Orthopedic surgery and anesthesia residents and orthopedic operating room nurses between the ages of 18-60 who do not have cardiological, neurological and psychiatric diseases, have had fluoroscopic operations lasting more than 2 hours, wear protective scopy gowns and collar during surgery
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate | In the perioperative period
  Pulse oximeter
Non Invasive Blood Pressure | In the perioperative period
  Syphgmomanometer
Weight | In the perioperative period
  Weighing machine

SECONDARY OUTCOMES:
Diarrhea | 2 hours after surgery
  Verbal answers
Visual Analog Scale (VAS) Score | 15 minutes after surgery
  VAS Score Scale (Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain(0 mm)" and "worst pain(100mm)".)
Radiation Exposure Time on Fluoroscopy Device | During surgery
  Chronometer
Rad Measurement | 5 minutes after surgery
  Personal Dosimeter
Total Time in the Operating Room | During surgery
  Chronometer
Mini Mental State Examination | 15 minutes after surgery
  Mini Mental State Examination Scale (This scale is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.)

CONTACTS AND LOCATIONS:
Overall Officials: Nur Canbolat, MD, Principal Investigator — Istanbul University Faculty of Medicine Department of Anesthesiology; Elif Aygün, MD, Principal Investigator — Istanbul University Faculty of Medicine Department of Anesthesiology; Cansu Uzunturk, MD, Principal Investigator — Istanbul University Faculty of Medicine Department of Anesthesiology; Evren Aygun, MD, Study Director — Istanbul University Faculty of Medicine Department of Anesthesiology; Yavuz Saglam, MD, Study Chair — Istanbul University Faculty of Medicine Department of Orthopedics; Mehmet I Buget, Assoc. Prof., Study Chair — Istanbul University Faculty of Medicine Department of Anesthesiology
Locations (1):
- Istanbul University, Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohsen S, Elham H, Hassan V, Sajad B, Mohammad G, Razieh R (2016) Hematological findings in medical professionals involved at intraoperative fluoroscopy. Glob J Health Sci 8:12
- [Background] Sailer AM, Vergoossen L, Paulis L, van Zwam WH, Das M, Wildberger JE, Jeukens CRLPN. Personalized Feedback on Staff Dose in Fluoroscopy-Guided Interventions: A New Era in Radiation Dose Monitoring. Cardiovasc Intervent Radiol. 2017 Nov;40(11):1756-1762. doi: 10.1007/s00270-017-1690-5. Epub 2017 May 12. PMID 28500459